CLINICAL TRIAL: NCT01600469
Title: NMDA-enhancing Agent for Treatment of Mild Cognitive Impairment and Mild Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99-2452A3
Record Dates: First submitted 2012-05-14; First posted 2012-05-17 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2011-04

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Alzheimer's disease; mild cognitive impairment; NMDA
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAOI-B (Experimental)
  Interventions: Drug: DAOI-B
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DAOI-B — 250-1500 mg/day, oral, for 24 weeks
  Arms: DAOI-B
Other: Placebo — placebo, oral, for 24 weeks
  Arms: Placebo

SUMMARY:
NMDA activation plays an important role in learning and memory. NMDA receptors were found to decrease in the frontal lobe and hippocampus of Alzheimer's disease and mild cognitive function impairment. This study is a randomized, double-blind, placebo-controlled drug trial. All patients will be allocated randomly to 2 groups: (1) NMDA enhancer: DAOI-B group (starting dose: 250-500 mg/d); (2) placebo group. The study period is 24 weeks. The investigators hypothesize that DAOI-B may yield better efficacy than placebo for cognitive function in patients with mild cognitive impairment or mild Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild cognitive impairment or mild Alzheimer's
* MMSE between 17-26
* CDR 0.5 or 1

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* substance abuse/dependence
* Parkinson disease
* epilepsy
* major depressive disorder
* dementia with psychotic features
* major physical illnesses
* severe visual or hearing impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Alzheimer's disease assessment scale-cognitive subscale in week 8, 16 and 24 | Week 0, 8, 16, 24

SECONDARY OUTCOMES:
Change from baseline in Mini Mental Status Examination at week 8, 16 and 24 | Week 0, 8, 16, 24
Change from baseline in Instrumental Activities of Daily Living at week 8, 16 and 24 | Week 0, 8, 16, 24
Change from baseline in Verbal learning and memory at week 24 | Week 0, 24
Change from baseline in Digit Span subtest of the Wechsler Memory Scale at week 24 | Week 0, 24

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-yuan Lane, MD, PhD, Study Chair — Departments of Psychiatry, China Medical University Hospital, Taichung, Taiwan
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung, Taiwan, Taiwan